CLINICAL TRIAL: NCT00787189
Title: The Effects of the Erchonia Hearing Laser on Word Recognition in Hearing Impaired Individuals Clinical Study Protocol
Brief Title: Study of Low Level Laser Therapy and Word Recognition in Hearing Impaired Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHL-001
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Sensorineural Hearing Loss
Keywords: sensorineural hearing loss; tinnitus; word recognition
MeSH Terms: conditions — Hearing Loss, Sensorineural; Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Hearing Laser (Active Comparator): Active low level laser light therapy of 635 nanometers (nm)
  Interventions: Device: The Hearing Laser
- Placebo Laser (Placebo Comparator): inactive low level laser light therapy with no therapeutic output
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: The Hearing Laser — Two 6-minute low level laser light applications to the head/neck/ears region, each one week apart.
  Arms: The Hearing Laser
Device: Placebo Laser — inactive low level laser light therapy with no therapeutic output
  Arms: Placebo Laser

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of low level laser light therapy when applied around the head and ears in improving unaided word recognition in ears with sensorineural hearing loss.

DETAILED DESCRIPTION:
Sensorineural hearing loss accounts for about 90% of all hearing loss and is found in 23% of individuals older than 65 years. Sensorineural hearing loss occurs when the hair cells of the inner ear and the neural pathways to the auditory cortex are damaged. In most cases, sensorineural hearing loss cannot be improved, reversed or 'cured.' Current treatment options focus on methods that amplify external sounds and on teaching the patient various strategies to 'retrain' the brain to interpret external stimuli. Low Level Laser Therapy was first applied for the treatment of inner ear diseases by Uwe Witt, MD of Hamburg, Germany in the 1980's. Hearing impaired patients have inflammation and/or atrophy of the tissues and neural pathways connected to and supporting the cochlea's cilia hair structure, the hearing mechanism of the inner ear. Low level laser therapy is believed to stimulate the mitochondria of the adipocyte cells, which subsequently increases the production of ATP. The resultant surge in ATP production works to repair damaged tissue and regenerate cells reversing some of the damage incurred to the cochlea and thus improving aspects of hearing function.

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural hearing loss.
* Mild or greater degree.
* Adult onset.
* Gradual onset.
* Hearing loss stable over past 12 months.
* Etiology of presbyacusis or noise-induced hearing loss.
* Unaided word recognition score between 28% and 86%.
* English as primary spoken language.
* Willing and able to abstain from other treatments or medications to improve hearing ability.
* Willing and able to abstain from work or other activities that involve loud noise exposure.

Exclusion Criteria:

* Central auditory processing disorder.
* Active/recurrent middle ear infection.
* Meniere's disease.
* Tympanic membrane perforation/tubes.
* Cochlear implant.
* Removal of acoustic neuroma.
* Hyperacusis/misphonia.
* Photosensitivity disorder.
* Active infection/wound in head/ear region.
* Pregnant/lactating.
* Serious mental health illness.
* Significant developmental disability/cognitive impairment.
* History of drug/alcohol abuse.
* Involvement in litigation/worker's compensation/disability benefits for hearing loss.
* Other research participation in past 90 days.
* Use of ototoxic medications known to cause temporary or permanent hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty McNamara, M.S., CCC-A, Principal Investigator — Maryjane Rees Language Speech & Hearing Center
Locations (1):
- McDonald Hearing Centers, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 subjects (80 ears) were recruited across two hearing aid and evaluation test sites from May, 2007 to October, 2008.
Pre-assignment Details: 4 subjects (8 ears) were disqualified because the word recognition score recorded for study qualification purposes exceeded the upper inclusive limit of 86% words correct. 4 subjects (8 ears) were disqualified because the subject's primary spoken language was not English, which was also a study exclusion criteria.
Groups:
- Active: Active laser device
- Control: Placebo laser device
Period: Overall Study
Arm/Group | Active | Control
Started | 32 | 32
Completed | 30 (To study end point.) | 30 (To study end point.)
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 26 | 32 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.94 (5.92) | 76.00 (9.86) | 77.47 (8.265)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 22 | 14 | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants Whose Change in Percent Correct Word Recognition Scores From Baseline to One Week After Study Treatment Equalled or Exceeded the Minimum Change in a Reference Chart.
Description: Participants were asked to repeat 50 words presented one at a time through headphones to each ear separately at a comfortable listening level to the participant. The 50 words were from a phonetically-balanced list of monosyllabic words called the Central Institute for the Deaf (CID) W-22 lists. For each ear, each word repeated correctly was scored '1'. The total number correct for each ear was summed and multiplied by 2 to attain the percent of total words repeated correctly for each ear. The change in this percent from baseline to one week after study treatment was referenced against a chart. If the change was equal to or greater than the corresponding value in the chart, the participant was considered to have a successful study outcome.
Time Frame: baseline and one week
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 32 | 32
participants | 15 | 2
Statistical Analysis 1: Comparison: Active vs Control; Test type: Superiority or Other; p < 0.0005, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Active | Control
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No